CLINICAL TRIAL: NCT00583713
Title: An Open Label Study to Assess the Effect of BLI800 on Safety and Clinical Chemistry Parameters
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Russell Pelham, Ph.D., Braintree Laboratories, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLI-800-202
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-10

CONDITIONS: Colonoscopy; Bowel Preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Renal Group (Experimental): Patients with moderate renal impairment
  Interventions: Drug: BLI-800
- Healthy volunteers (Active Comparator): Healthy volunteers
  Interventions: Drug: BLI-800
- Hepatic Group (Experimental): Patients with mild/moderate hepatic impairment.
  Interventions: Drug: BLI-800

INTERVENTIONS:
Drug: BLI-800 — BLI-800 oral solution (two doses)

SUMMARY:
To evaluate and compare the effects on safety measures and clinical chemistry after BLI800 in two groups of patients and one group of healthy controls. The patient groups will be those with mild or moderate hepatic impairment or moderate renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female adults who are:

  * With Child-Pugh Hepatic Dysfunction Stage A or B, or
  * With Moderate Renal Disease or
  * Healthy subjects matched to those who are enrolled in this study
* Subjects who are considered to have only clinically non-significant conditions, as judged by the Principal Investigator and based on physical examination, laboratory profiles, medical history and ECG.
* Female subjects who are not surgically sterile (i.e., having had a hysterectomy, bilateral oophorectomy or tubal ligation) or who are not at least 2 years naturally postmenopausal must agree to use an acceptable form of contraception.
* Provide voluntary consent in writing to participate in this study.

Exclusion Criteria:

* Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or megacolon.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects who, in the opinion of the Principal Investigator, have uncontrolled clinically significant pre-existing electrolyte disturbances, based on the Screening visit laboratory results.
* Subjects with present or prior NYHA Functional Classification grade III or IV congestive heart failure.
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days.
* Subjects with a history of allergic or adverse response to any BLI-800 component.
* Subjects who donated more than one pint of blood within 30 days prior to the study.
* Subjects who donated plasma within 7 days prior to the study.
* Subjects who had an abnormal diet or substantial changes in eating habits within 30 days prior to the start of the study.
* Subjects who have had a bowel cleansing procedure within the past month or who have taken a laxative within the 5 days (120 hours) prior to dosing or who require a laxative every day.
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Pelham, Ph.D., Study Director — Braintree Laboratories, Inc.
Locations (1):
- Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Group: BLI-800 oral solution in patients with moderate renal impairment
- Healthy Volunteers: BLI-800 oral solution in healthy volunteers
- Hepatic Group: BLI-800 oral solution in patients with mild/moderate hepatic impairment.
Period: Overall Study
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 6 | 17
  >=65 years | 1 | 0 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 53.8 (7.96) | 49.0 (6.93) | 51.2 (5.74) | 51.3 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 3 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
µmol/L | 717.0 (270.84) | 499.5 (165.00) | 560.2 (152.75)

2. Secondary Outcome: Urinary Sulfate Concentration
Time Frame: pre-dose to 6 days post-dose
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
mg/dL
  Pre-dose 1 | 91.58 (40.12) | 131.20 (46.98) | 86.92 (50.09)
  Day 3 | 135.53 (86.28) | 145.62 (111.02) | 89.83 (67.81)
  Day 6 | 96.98 (47.61) | 134.65 (74.72) | 70.82 (83.64)

3. Primary Outcome: Time to Maximum Concentration
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
hours | 17.5 (2.95) | 16.8 (8.16) | 14.2 (5.00)

4. Primary Outcome: Terminal Half-life
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
hours | 10.16 (9.32) | 8.51 (4.57) | 5.58 (2.31)

5. Primary Outcome: Area Under the Curve for the 24-hour Dosing Interval
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: µmol*hr/L
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
µmol*hr/L | 12,332.95 (4,193.54) | 8,029.88 (3,424.42) | 10,751.75 (2,878.17)

6. Primary Outcome: Elimination Rate Constant
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Number analyzed (Participants) | 6 | 6 | 6
1/hr | 0.127 (0.09) | 0.107 (0.06) | 0.141 (0.050)

ADVERSE EVENTS:
Arm/Group | Renal Group | Healthy Volunteers | Hepatic Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Group (N=6) | Healthy Volunteers (N=6) | Hepatic Group (N=6)
Abdominal cramping (Gastrointestinal disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 3 | 3
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Emesis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Perianal irritation (Gastrointestinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abnormal urinalysis (Investigations) | 0 | 0 | 1
Elevated serum creatinine (Investigations) | 0 | 1 | 1
Symptomatic hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other